CLINICAL TRIAL: NCT04494009
Title: Randomized Phase II Trial of a PD-1 Inhibitor INCMGA00012 as Consolidation Therapy After Definitive Concurrent Chemoradiotherapy for Patients With Locally Advanced Esophageal Squamous Cell Carcinoma (RHAPSODY)
Brief Title: PD-1 Inhibitor INCMGA00012 as Consolidation Therapy After Definitive Concurrent Chemoradiotherapy
Acronym: RHAPSODY
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sook Ryun Park, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MC20-01
Record Dates: First submitted 2020-07-14; First posted 2020-07-31 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- INCMGA00012 군 (Experimental): INCMGA00012 500 mg iv every 4 weeks for up to 12 months
  Interventions: Drug: INCMGA00012
- Observation arm (No Intervention): followed up every 12 weeks for up to 12 months

INTERVENTIONS:
Drug: INCMGA00012 — INCMGA00012 (also known as MGA012) is a humanized, hinge-stabilized IgG4 monoclonal antibody against human PD-1, which blocks the interaction of PD-1 with PD-L1 and PD-L2, interrupting PD-1 signaling, enhances antigen-induced interferon-γ release, and has a favorable preclinical profile.
  Arms: INCMGA00012 군

SUMMARY:
This study is a randomized, multi-center, open-label, phase II study of a PD-1 inhibitor (INCMGA00012) versus observation as consolidation therapy after definitive concurrent chemoradiotherapy in patients with locally advanced ESCC who have not progressed following definitive chemoradiotherapy.

DETAILED DESCRIPTION:
This study is a randomized, multi-center, open-label, phase II study of a PD-1 inhibitor (INCMGA00012) versus observation as consolidation therapy after definitive concurrent chemoradiotherapy in patients with locally advanced ESCC who have not progressed following definitive chemoradiotherapy.

Patients must have received definitive concurrent chemoradiotherapy for locally advanced ESCC (cT1b N1-3 M0 or T2-4b N0-3 M0 according to the 8th American Joint Committee on Cancer [AJCC] staging system) because of unresectable disease status (such as cervical esophageal cancer and cTb), medically inoperable status, or patient's refusal of undergoing surgery.

Patients must not have progressed following definitive chemoradiotherapy consisting of fluoropyrimidine or taxane plus platinum chemotherapy (including, but not limited to fluorouracil plus cisplatin, capecitabine plus cisplatin, and paclitaxel plus carboplatin according to the institute standard of care regimens) concurrent with radiation therapy (a total dose of at least 50 Gy). One or two cycles of induction chemotherapy before chemoradiotherapy is allowed, but chemotherapy after concurrent chemoradiotherapy is not allowed.

Approximately 110 patients who have not progressed following definitive chemoradiotherapy for locally advanced ESCC will be randomly assigned within 4-8 weeks after completing chemoradiotherapy in a 1:1 ratio to the INCMGA00012 arm or observation arm.

* INCMGA00012 arm (500 mg iv every 4 weeks for up to 12 months)
* Observation arm (followed-up every 3 months) Randomization will be stratified by Eastern Cooperative Oncology Group (ECOG) performance status (0-1 vs. 2), clinical response to definitive chemoradiation (complete response [CR] vs. non-CR), and institute.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial.
2. Be ≥19 years of age on the day of signing the informed consent.
3. Have ECOG performance status 0-2 (Appendix 1).
4. Have histologically proven esophageal squamous cell carcinoma (ESCC).
5. Have demonstrated cT1b N1-3 M0 or T2-4b N0-3 M0 (8th AJCC staging system) before definitive chemoradiotherapy (Appendix 2).
6. Have completed definitive concurrent chemoradiotherapy for esophageal cancer due to unresectable disease status (such as cervical esophageal cancer and T4b), medically inoperable status, or patient's refusal of undergoing surgery.
7. Have received fluoropyrimidine or taxane plus platinum chemotherapy (including, but not limited to fluorouracil plus cisplatin, capecitabine plus cisplatin, and paclitaxel plus carboplatin according to the institute standard of care regimens) concurrent with radiation therapy. One or two cycles of induction chemotherapy before chemoradiotherapy is allowed, but chemotherapy after concurrent chemoradiotherapy is not allowed.
8. Have received a total dose of radiation of at least 50 Gy as part of concurrent chemoradiotherapy.
9. Have not progressed following definitive chemoradiotherapy assessed by 18F-FDG-PET (or PET-CT) scan, esophagogastroduodenoscopy (EGD), and chest CT. Clinical response should be evaluated within 4 to 8 weeks after completing definitive chemoradiotherapy, and within 3 weeks before randomization.
10. Have available pre-treatment tumor tissue for biomarker analyses. Either 1 formalin-fixed paraffin embedded (FFPE) tumor tissue block or 20 unstained tumor tissue slides must be submitted for biomarker evaluation. Post-chemoradiation biopsy should be performed if it is technically feasible and is not associated with unacceptable clinical risk, and in case of pathologic residual cancer, tumor tissue for biomarker analyses should be submitted (Either 1 FFPE tumor tissue block or 20 unstained tumor tissue slides).
11. Have adequate major organ functions as demonstrated by following laboratory results obtained within 14 days prior to randomization (these lab criteria should be also met within 7 days before initiation of study drug):

    * Adequate bone marrow function as defined by absolute neutrophil count (ANC) ≥ 1,000/mm3 and platelet count ≥ 75,000/mm3 without receiving growth factors or blood transfusion within 7 days before the laboratory testing.
    * Adequate renal function with serum creatinine ≤ 1.5 x upper limit of normal (ULN) or creatinine clearance ≥50 mL/minute by calculation using the Cockcroft-Gault formula (Appendix 3) or measurement using a preferred method per institute standard of care.
    * Adequate hepatic function with alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN, and serum total bilirubin ≤ 1.5 x ULN except for subjects with Gilbert syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology) who may be enrolled despite a total bilirubin level > 1.5 x ULN.
12. Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 14 days prior to randomization. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
13. Female subjects of childbearing potential randomized to the INCMGA00012 arm must be willing to use an adequate method of contraception for the duration of study treatment and 90 days after the last dose of study treatment.
14. Non-sterile male subjects randomized to the INCMGA00012 arm and who have female sexual partner(s) of childbearing potential must agree to use an adequate method of contraception for the duration of study treatment and 90 days after the last dose of study treatment.

Exclusion Criteria:

1. Has demonstrated disease progression while or after completion of definitive chemoradiotherapy for locally advanced ESCC.
2. Has received sequential chemotherapy or chemoradiotherapy after completion of concurrent chemoradiotherapy for locally advanced ESCC.
3. Has received any immunotherapy or investigational drug within 4 weeks prior to randomization.
4. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
5. Any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy, investigational agent, or local treatment (except for stent insertion or feeding enterostomy for palliative intent) for cancer treatment.
6. Any unresolved toxicities CTCAE grade ≥2 from prior therapy with the exception of alopecia, fatigue, and neuropathy.
7. Has undergone major surgery within 4 weeks prior to entry into the study.
8. Has an active autoimmune disease that has required systemic treatment within the 2 years prior to entry into the study (i.e., with use of disease-modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal insufficiency of pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
9. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
10. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (>10 mg/day prednisolone or equivalents) or any other form of immunosuppressive therapy within 14 days prior to entry into the study. Note: A use of topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption) is allowed. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
11. Has a history of organ transplant, including stem cell allograft.
12. Has received a live vaccine within 30 days prior to entry into the study. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
13. Has an active infection requiring systemic therapy.
14. Has known history of Human Immunodeficiency Virus (HIV) infection.
15. Has active HBV (detectable HBsAg or HBV DNA) or HCV infection (detectable HCV RNA):

    o For the subject receiving antiviral agents for HBV at screening, if the subject has been treated for > 2 weeks and HBV DNA is <500 IU/mL (or 2,500 copies/mL) prior to randomization, the subject will be allowed to be enrolled in the study. Antiviral agent should be continued for 6 months after study drug treatment discontinuation.
16. Has known history of, or any evidence of interstitial lung disease, non-infectious pneumonitis, or pulmonary fibrosis diagnosed based on imaging or clinical findings. Note: Subjects with radiation pneumonitis may be enrolled if the radiation pneumonitis has been confirmed as stable (beyond acute phase) and is unlikely to recur.
17. Has history of another primary malignancy requiring active treatment within the previous 3 years except for adequately treated basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ (e.g., of cervix, breast, prostate).
18. Has medical or psychiatric conditions that compromise the subject's ability to give informed consent or to complete the protocol or a history of non-compliance.
19. Has significant cardiovascular impairment within 6 months prior to entry to the study such as history of congestive heart failure meeting New York Heart Association (NYHA) Class III or IV, unstable angina, myocardial infarction, cerebrovascular accident, or cardiac arrhythmia associated with hemodynamic instability.
20. Has a history of severe hypersensitivity to antibody products.
21. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
22. Is a pregnant or breastfeeding woman.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-09-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival per RECIST 1.1 | 5 Years
  Every 12 weeks during the first two years after randomization then every 24 weeks

SECONDARY OUTCOMES:
Overall Survival | 5 Years
  every visit
Progression Free Survival per iRECIST | 5 Years
  Every 12 weeks during the first two years after randomization then every 24 weeks
Time To Progression per RECIST 1.1 | 5 Years
  Every 12 weeks during the first two years after randomization then every 24 weeks
Time To Progression per iRECIST Time To Progression per iRECIST | 5 Years
  Every 12 weeks during the first two years after randomization then every 24 weeks
To compare pattern of first cause of progression | 5 Years
  Every 12 weeks during the first two years after randomization then every 24 weeks
To compare the safety and tolerability(NCI-CTCAE version 5.0) | 5 Years
  every visit
HRQoL, time to deterioration | 5 Years
  Every 12 weeks during the first two years after randomization then every 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sook Ryun Park, MD, Ph.D., Study Chair — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chitti B, Pham A, Marcott S, Wang X, Potters L, Wernicke AG, Parashar B. Temporal Changes in Esophageal Cancer Mortality by Geographic Region: A Population-based Analysis. Cureus. 2018 Nov 15;10(11):e3596. doi: 10.7759/cureus.3596. PMID 30680257
- [Background] Murphy G, McCormack V, Abedi-Ardekani B, Arnold M, Camargo MC, Dar NA, Dawsey SM, Etemadi A, Fitzgerald RC, Fleischer DE, Freedman ND, Goldstein AM, Gopal S, Hashemian M, Hu N, Hyland PL, Kaimila B, Kamangar F, Malekzadeh R, Mathew CG, Menya D, Mulima G, Mwachiro MM, Mwasamwaja A, Pritchett N, Qiao YL, Ribeiro-Pinto LF, Ricciardone M, Schuz J, Sitas F, Taylor PR, Van Loon K, Wang SM, Wei WQ, Wild CP, Wu C, Abnet CC, Chanock SJ, Brennan P. International cancer seminars: a focus on esophageal squamous cell carcinoma. Ann Oncol. 2017 Sep 1;28(9):2086-2093. doi: 10.1093/annonc/mdx279. PMID 28911061